CLINICAL TRIAL: NCT03013608
Title: Children's Nail Bed Injuries : Study of the Efficacy of the Simple Relocation of Nail Plate
Acronym: Ongl'HUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6529
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2019-08

CONDITIONS: Nail Bed Injury
Keywords: Nail bed injury; Nail bed injuries; Nail; Children; Fingertip injury
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- relocation of nail plate (Experimental): the simple relocation of the nail plate in nailbed injuries in paediatric population
  Interventions: Procedure: Simple relocation of the nail plate in nailbed injuries in paediatric population

INTERVENTIONS:
Procedure: Simple relocation of the nail plate in nailbed injuries in paediatric population — Repositioning the nail bed without sutures
  Other Names: Reparation of the nail bed injuries; Repositioning the nail bed without sutures; Relocation of the nail

SUMMARY:
Nail bed injuries in children, most frequently under 3 years-old, result in crush injuries. The frequency is around 34 percent of the children hand injuries (Claudet et al, 2007). The empirical reparation technique is the nail bed suture and the relocation of the nail plate. However, some authors think that suture the nail bed could increase the traumatism of the nail bed because of the needle, the crush by the clamps and by the stitches too tight (Langlois, Yam). An author has proposed, in a prospective, randomized clinical trial to treat the nail bed injuries with a glue: the 2-octylcyanoacrylate, without suture of the nail bed. Advantages of this technique, claimed by the author, was time saving, with an aesthetical result as same as the treatment with suture of the nail bed. A same study validated the technique in a paediatric population (Langlois et al., 2010). So, it seems that it is not necessary to suture the nail bed. But, in our practice, the investigators noted complications not mentioned in previous studies: hematomas causing pain, effusion and dislocation of the nail plate, with constrain the patient to consult in emergency. The 2-octylcyanoacrylate is difficult to use in nail bed injuries and is expensive. Our hypothesis is the simple relocation of the nail plate in nail bed injuries in paediatric population is enough to have good to excellent aesthetical results, with less complications and a lower cost, than the other techniques. The aim of this study is to assess the aesthetical results 3 months after simple relocation of the nail plate for nail bed injuries in children.

ELIGIBILITY:
Inclusion Criteria:

* age under 18 yo
* nail bed injuries and/or nail matrix
* nail plate > 30% of the surface comparing the opposite side
* one or more digits
* signature of the 2 parents
* social security

Exclusion Criteria:

* loss of more than 30% of the surface of the nail bed
* Multiples lesions: nerve injury, tendon, fracture or luxation without indication of osteosynthesis, loss of skin with indication of a flap
* osteosynthesis of the distal phalanx
* injuries by bite
* previous pathology of the nail
* contraindication of Lidocaine, bicarbonate de sodium, Kalinox, Biseptine, Vicryl rapide, Adaptic
* no information possible
* pregnancy
* breastfeeding
* other inclusion in another study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Nail aesthetical results | The evaluation is assessed at 6 months after the treatmen6
  Evaluation with the Zook's scale at 6 months postoperative based on photographs of the injured finger compared with the finger on the opposite side. The evaluation will be done by five persons (surgeons, nurses, therapists….)

SECONDARY OUTCOMES:
Complications rate at short term (before 15 days): haematoma, infection, dislocation of the nail plate,: hook nail | at 15 days
The pain with an analogic scale for children over 7 years-old, | at 6 months
Satisfaction rate at 6 months, compared with the contralateral finger, by the children (if possible) and by parents, on a scale to 0 (not satisfied) to 10 (very satisfied). | at 6 months
  photographs, evaluation of the roughness by the surgeon, the nurse and parents, satisfaction of the aspect of the nail on a scale (0 to 10)
Complications rate: haematoma, infection, dislocation of the nail plate,at medium term (between 15 days and 3 months): hook nail | at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Strasbourg,, Strasbourg, France